CLINICAL TRIAL: NCT04937569
Title: Ivermectin Versus Standard Treatment in Mild COVID-19: a Prospective Cohort Study.
Brief Title: Ivermectin Versus Standard Treatment in Mild COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU-Ivercom
Record Dates: First submitted 2021-06-23; First posted 2021-06-24 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; Ivermectin; Standard therapy; ICU admission; Clinical improvement; Side effects; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Ivermectin + standard treatment (Active Comparator): Patients will receive 4-days course of Ivermectin 400 microgram/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast plus standard treatment (Azithromycin 500mg once daily for 5 days, Paracetamol 500mg every 8 hours, vitamin C 1gm once daily, Zinc 50 mg once daily, Lactoferrin 100mg sachets twice daily and prophylactic or therapeutic anticoagulation if D-dimer is elevated.
  Interventions: Drug: Ivermectin Tablets
- Group-2: Standard treatment only (Other): This group will receive the standard treatment protocol as outlined above according to the Egyptian Ministry of Health protocol of treating cases with mild COVID-19.
  Interventions: Drug: Ivermectin Tablets

INTERVENTIONS:
Drug: Ivermectin Tablets — 4-days course of Ivermectin 400 microgram/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast

SUMMARY:
Rationale: Ivermectin, an inexpensive and available antiparasitic drug, with favourable safety profile, showed inhibitory effect on SARS-CoV2 viral replication in-vitro and in animal models. Several research groups investigated Ivermectin in COVID-19, particularly in mild symptomatic disease. There is high degree of uncertainty on its effects on clinical outcomes and larger studies are needed.

Objectives: Plan to study the effect of Ivermectin versus standard treatment in patients with confirmed mild COVID-19.

Study design: Multi-centre prospective cohort study Settings: Assiut University Hospital (Assiut University), Aswan and others, Egypt.

Study Population: Patients with confirmed mild COVID-19. Intervention: Patients with mild symptomatic COVID-19 attending the participating out-patient clinics in different centers will receive either Ivermectin + Standard treatment or Standard treatment only. All new mild symptomatic COVID-19 patients will receive Ivermectin + Standard treatment for the first two weeks of the study. During the following four weeks, all new patients will receive standard treatment only. These cycles will be repeated until 822 patients are recruited in each arm. Patients assigned to Ivermectin + Standard treatment or standard treatment only will remain as such throughout the study and during the follow- up period.

Primary outcome measures: The primary outcome will be rate of intensive care admission.

Secondary outcome measures: Secondary outcomes will be time to clinical improvement, the clinical state using 7-point ordinal scale at different time points, need for home oxygenation, hospitalization, hospital supplemental oxygen >24 hours, Non- invasive ventilation ( High- flow nasal cannula, High- velocity nasal insufflation or BiPAP), duration of hospitalization, duration of ICU stay and deaths within 21 days,.

Power calculation:

With a prospective cohort design, a sample size of 822 cases per group is estimated (1644 for the whole study). This calculation depends on a rate of ICU admission in mild symptomatic COVID-19 cases of 8.5%, an assumption that Ivermectin can reduce this rate by 50%, at a study power of 80%, and confidence limit of 0.95.

DETAILED DESCRIPTION:
1. Introduction and rationale: An outbreak of atypical pneumonia of unknown cause erupted in Wuhan, China in December 2019. The symptoms ranged from mild symptoms to severe acute respiratory distress syndrome, with multi-organ affection leading to patients' death. Within few weeks, genetic sequence of the causative virus was identified to be close to Severe Acute Respiratory Distress Virus (SARS-CoV) (Zhou et al, 2020). The newly identified virus was named Novel Coronavirus or SARS-CoV2, and the clinical disease as COVID-19 (Chung et al, 2021). The disease spread rapidly with travel movements around the world and the World Health organization announced the COVID-19 as a pandemic on March 11th, 2020 (Cucinotta and Vanelli, 2020). The worldwide disease toll approached more the 165 million confirmed cases including more than 3.5 million deaths as of May 21st, 2021, making it the worst pandemic in the last 100 years [WHO Coronavirus (COVID-19) Dashboard].

Attempting to find therapeutic options for COVID-19, viral inhibitor drugs that have been used against influenza and HIV, were repurposed to be tested against SARS-CoV2. These include Chloroquine/ Hydroxychloroquine which inhibit viral entry and endocytosis in vitro, protease inhibitors Lopinavir-Ritonavir which disrupt viral replication in-vitro, and RNA dependent polymerase inhibitors including Ribavirin, Favipiravir and Remdesivir (Wiersinga et al, 2020). Only Remdesivir showed initial promising results in a randomized clinical trial (Beigel et al, 2020), however, currently the World Health Organization recommends against its use in any disease severity (Lamontage et al, 2021).

Ivermectin is an inexpensive and available antiparasitic drug, with favourable safety profile. It showed inhibitory effect on SARS-CoV2 viral replication in vitro and in animal models (Formiga et al, 2021). Several research groups investigated Ivermectin in COVID-19, particularly early in mild disease where viral replication is more active (Kory et al, 2021). In its living guideline on drugs used to treat COVID-19, the WHO recommended against the use of Ivermectin in COVID-19, regardless of duration of symptoms or disease severity, except in the contest of clinical trials. The reason was high degree of uncertainty about clinical outcomes of importance to the patients like time to clinical improvement, hospital admission, duration of hospitalization, mechanical ventilation and mortality. The WHO recommends larger and well-designed studies to solve this uncertainty (Lamontage et al, 2021).

In the present study protocol, the investigators plan to study the effect of Ivermectin versus standard treatment in patients with confirmed mild symptomatic COVID-19. The primary outcome will be rate of intensive care admission. Secondary outcomes will be time to clinical improvement, patient's clinical state using 7-point ordinal scale at different time points, proportion of subjects needing hospitalization, supplemental oxygen >24 hours, duration of hospitalization, duration of ICU stay or death within 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed mild cases of COVID-19 defined as: symptomatic patients with any of COVID-19 symptoms (fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell),
* In addition to absolute leucopoenia (< 4000) / absolute lymphopenia (< 1000), positive CRP (C-reactive protein), high serum ferritin and/or positive PCR for SARS-CoV-2 in nasopharyngeal swab.
* no dyspnea and no abnormalities on high resolution chest imaging (HRCT).
* Patients should be at home (not admitted to hospital) with no supplemental oxygen treatment.

Exclusion Criteria:

* • Asymptomatic patients

  * Dyspnoea or abnormalities on chest imaging
  * Hospital admission
  * Severe pneumonia
  * Impairment in liver functions
  * Received Ivermection in the last 5 days before being included in the study.
  * Pregnancy is an exclusion criterion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1644 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of ICU admission in mild COVID-19 cases | 21 days
  Indications of ICU admission, Respiratory rate (RR) > 30 cycle/min, Oxygen saturation < 92% at room air, PaO2/FiO2 ratio < 300, Chest radiography showing more than 50% lung lesions, or progressive lesions within 24-48 hours, Critically ill if RR > 30, Oxygen saturation < 92%, or PaO2/FiO2 ratio < 200 despite oxygen therapy.

SECONDARY OUTCOMES:
Time to clinical improvement. | 21 days
  days to fever, dyspnea, cough improvement
Overall clinical state, using the 7-point ordinal scale | 21 days
  7-point ordinal scale is: 1. Death 2. Hospitalized, on invasive mechanical ventilation or Extracorporeal Membrane Oxygenation 3. Hospitalized, on non-invasive ventilation or high flow oxygen 4. Hospitalized, requiring low flow supplemental oxygen 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise) 6. Hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care 7. Not hospitalized.
The duration of critical care interventions in each arm of the study. | 21 Days
  * The duration of supplemental oxygen in each arm of the study.
  * The duration of hospitalization in each arm of the study.
  * The duration of stay in the ICU in each arm of the study.
• Proportion of subjects who develop adverse events associated with the study drug. | 21 days
  percentage of patients having SE as headache, dizziness, diarrhoea, nausea, disturbed vision, tremors, skin discoloration, skin rash, swelling, vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Aliae AR Mohamed-Hussein, MD, Principal Investigator — Assiut University; Essam R Othman, MD, Study Director — Assiut University; Ben WJ Mol, MD, Study Chair — Monash University
Locations (1):
- Aliae AR Mohamed-Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No